CLINICAL TRIAL: NCT01094496
Title: A Phase II, Open-Label Study of the CDX-1307 Vaccine Regimen as Neoadjuvant and Adjuvant Therapy in Patients With Newly Diagnosed Muscle-Invasive Bladder Cancer Expressing hCG-β
Brief Title: A Study of the CDX-1307 Vaccine Regimen in Patients With Newly Diagnosed Muscle-Invasive Bladder Cancer (The "N-ABLE" Study)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Portfolio prioritization due to slow enrollment
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX1307-03
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2016-02

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; immunotherapy; cystectomy; cancer vaccine; human chorionic gonadotropin; hCG; urogenital neoplasms; urinary bladder neoplasms; muscle invasive; non-metastatic; transitional cell (urothelial) bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urogenital Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CDX-1307 Vaccine Regimen (Experimental): Chemotherapy with CDX-1307 vaccine regimen (neoadjuvant phase), followed by bladder removal surgery (cystectomy). CDX-1307 vaccine regimen will continue to be given for up-to 1 year post-surgery (adjuvant/long-term follow-up phase).
  Interventions: Biological: CDX-1307 Vaccine Regimen; Drug: Chemotherapy

INTERVENTIONS:
Biological: CDX-1307 Vaccine Regimen — CDX-1307 vaccine co-administered with immune adjuvants (GM-CSF, Poly-ICLC and Resiquimod)
Drug: Chemotherapy

SUMMARY:
The major purpose of this study is to examine the anti-tumor activity of the CDX-1307 vaccine regimen when it is given before and after bladder cancer surgery. The study will also provide information about the safety of the vaccine regimen when given in combination with chemotherapy, and how it affects the immune systems.

DETAILED DESCRIPTION:
CDX-1307 is an experimental vaccine that is designed to generate an immune response against a protein called human chorionic gonadotropin-beta (hCG-β). hCG-β is made by several types of cancers, including bladder cancer, and has been shown to be associated with shorter times to development of metastases and reduced survival in bladder cancer. In this study, it is hoped that administering the CDX-1307 vaccine will cause the body's immune system to attack bladder cancer cells in order to kill them or otherwise keep them from spreading or coming back.

Standard treatment for early stage, muscle invasive bladder cancer includes the administration of chemotherapy to shrink the tumor followed by surgical removal of the bladder (cystectomy).

This study will compare the effect of adding CDX-1307 administration to this standard treatment. CDX-1307 will be given with 3 different immune stimulants to try to increase the immune response against the tumor cells; collectively, this is called the "CDX-1307 vaccine regimen."

Only patients whose tumors make the hCG-β protein will be included in this study. Eligible patients will receive "standard of care" chemotherapy with the CDX-1307 vaccine regimen before surgery, and then CDX-1307 vaccine regimen alone (without chemotherapy) after surgery.

ELIGIBILITY:
Inclusion Criteria:

Among other criteria, patients must meet all of the following conditions to be eligible to be in the study:

1. 18 years of age or older.
2. Newly diagnosed muscle-invasive transitional cell (urothelial) bladder cancer where neoadjuvant chemotherapy and radical cystectomy with curative intent are indicated (i.e., American Joint Committee on Cancer (AJCC) stage T2-4a, Nany, M0). Patients must be entered into the study within eight weeks of their most recent diagnostic procedure, which is usually a diagnostic biopsy or transurethral resection of bladder tumor (TURBT) procedure.
3. Histopathologically confirmed, transitional cell (urothelial) carcinoma. Urothelial tumors with mixed histology (but with <50% variant) are eligible.
4. Tumor tissue (obtained during a prior procedure) confirmed to express hCG-β by a central laboratory.
5. Candidate for therapy with neoadjuvant chemotherapy.

Exclusion Criteria:

Among other criteria, patients who meet any of the following conditions are NOT eligible to be in the study:

1. Previous systemic chemotherapy or radiation for bladder cancer. Note: Prior immunotherapy or intravesical (administered within the bladder) chemotherapy for superficial disease is acceptable.
2. History of anaphylactic reaction following exposure to humanized or human therapeutic monoclonal antibodies, hypersensitivity to GM-CSF or yeast derived products, clinically meaningful allergic reactions to imiquimod, resiquimod, or any known hypersensitivity or prior reaction to any of the formulation excipients in the study drugs.
3. Concurrent chronic treatment with immunosuppressive or immunomodulatory agents, including any systemic steroid (exception: inhaled or topically applied steroids, and acute and chronic standard dose NSAIDs, are permitted).
4. Known infection with HIV, HBV or HCV.
5. Any underlying medical condition that, in the Investigator's opinion, will make the administration of study vaccine hazardous to the patient, would obscure the interpretation of adverse events, or would contraindicate receipt of neoadjuvant chemotherapy or surgical resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
2 year Recurrence-Free Survival Rate | 2 years following enrollment
  The 2-year recurrence-free survival rate will be estimated based on the proportion of patients who are classified as alive and without documented disease recurrence at this time point.
Duration of Recurrence-Free Survival | Up-to 4 years after bladder removal surgery (cystectomy)
  The duration of recurrence-free survival is defined as the number of months from enrollment to the earlier of disease recurrence or death (whatever the cause).

SECONDARY OUTCOMES:
Tumor response to neoadjuvant chemotherapy | At cystectomy (anticipated to be about 4 months post-enrollment)
  The tumor response to neoadjuvant chemotherapy will be evaluated as the proportion of patients who achieve a radiographic response as defined by the Response Evaluation Criteria for Solid Tumors (RECIST 1.1) or a pathologic complete response at cystectomy.
Overall survival | Up-to 4 years following bladder removal surgery (cystecomy)
  Overall survival is defined as the number of months from enrollment to the date of death (whatever the cause).
Safety / Tolerability | Through completion of study treatment (about 1 year post-resection)
  The number and percentage of patients experiencing one or more adverse events will be summarized by relationship to study drug and severity. Separate tabulations will be provided for the neoadjuvant and adjuvant treatment phases.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - BCG Oncology, PC, Phoenix, Arizona
  - University of California - San Diego, La Jolla, California
  - University of Southern California Norris Comprehensive Cancer Center LA-USC Medical Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky Markey Cancer Center Clinical Research Organization, Lexington, Kentucky
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Center, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Syracuse VA Medical Center, Syracuse, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania